CLINICAL TRIAL: NCT05248087
Title: Assessment of Patient-centered Outcomes Associated With the Expansion of Skeletally Constricted Upper Jaw in the Adolescents Using Two Types of Expanders: A Randomized Controlled Trial
Brief Title: Pain, Discomfort, and Functional Impairments During Maxillary Expansion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UDDS-Ortho-02-2022
Record Dates: First submitted 2022-02-10; First posted 2022-02-21 (Actual); Last update posted 2022-02-21 (Actual); Status verified 2022-02

CONDITIONS: Constriction
Keywords: Pain; Discomfort; Crossbite; Maxillary expansion
MeSH Terms: conditions — Constriction, Pathologic; Pain; Malocclusion

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The rapid maxillary expansion (Experimental): The rapid maxillary expansion will be applied using a McNamara-type (bonded) appliance.
  Interventions: Device: The bonded McNamara-type appliance
- The slow maxillary expansion (Active Comparator): The slow maxillary expansion will be applied using a removable palatal expansion appliance.
  Interventions: Device: The removable palatal expansion appliance

INTERVENTIONS:
Device: The bonded McNamara-type appliance — The patient will be asked to expand twice a day until obtaining an overcorrection of 2-3 mm. Then the expander will be kept in place for three months as a retention period.
  Arms: The rapid maxillary expansion
Device: The removable palatal expansion appliance — The slow maxillary expansion will be applied using a removable palatal expansion appliance with a midline screw. The patient will be asked to expand twice a week until obtaining an overcorrection of 2-3 mm.
  Arms: The slow maxillary expansion

SUMMARY:
Maxillary expansion is associated with varying degrees of pain and functional impairments. The current study aims to compare rapid maxillary expansion using a McNamara-type (bonded) appliance and slow maxillary expansion using a removable palatal expansion appliance concerning patient-centered outcomes. Those outcomes will include pain and discomfort, mastication difficulties, swallowing difficulties, and pressure on the soft tissues.

DETAILED DESCRIPTION:
Skeletal maxillary constriction is one of the common orthodontic problems of all ages, which could be unilateral or bilateral. If it is neglected and not treated, it may result in later orthodontic problems such as skeletal deviation of the lower jaw. The current study aims to use two types of expanders to treat skeletal maxillary constriction in adolescents aged between 12 and 16 years. The study sample will include 52 patients who will be equally divided into two groups: the slow and the rapid maxillary expansion groups. Patients will be asked to answer a questionnaire within five assessment times during the expansion procedure. The questionnaire will contain four questions: 1) What is the degree of discomfort/pain? 2) What is the degree of mastication difficulties? 3) What is the degree of swallowing difficulties? 4) What is the degree of any sense of pressure in soft tissue?

ELIGIBILITY:
Inclusion Criteria:

1. Adolescents between 12 and 16 years.
2. Early permanent dentition.
3. Skeletal bilateral maxillary constriction.
4. There is no loss or absence of any permanent teeth except for the third molar.
5. Dental and skeletal class I/II malocclusion.
6. Normal/mild vertical growth pattern.

Exclusion Criteria:

1. Previous orthodontic treatment.
2. A severe horizontal growth pattern.
3. Any periodontal diseases.
4. Any general diseases or syndromes.

Ages: 12 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 52 (Actual)
Dates: Start 2020-02-20 (Actual); Primary Completion 2021-03-20 (Actual); Study Completion 2021-07-25 (Actual)

PRIMARY OUTCOMES:
Change in the levels of discomfort or pain | T1: after 24 hours; T2: on the 7th day; T3: on the 15th day; T4: after 1 month; T5: after 4 months
  The degree of pain and discomfort that patients feel will be determined using their answers to the following question (question 01):
  'What is the degree of discomfort/pain?' The Visual Analogue Scale (VAS) will be adopted to measure the degree of discomfort/pain.
Change in the levels of mastication difficulties | T1: after 24 hours; T2: on the 7th day; T3: on the 15th day; T4: after 1 month; T5: after 4 months
  The degree of mastication difficulties that patients feel will be determined using their answers to the following question (question 02):
  'What is the degree of mastication difficulties?' The Visual Analogue Scale (VAS) will be adopted to measure the degree of mastication difficulties.
Change in the levels of swallowing difficulties | T1: after 24 hours; T2: on the 7th day; T3: on the 15th day; T4: after 1 month; T5: after 4 months
  The degree of swallowing difficulties that patients feel will be determined using their answers to the following question (question 03):
  ' What is the degree of swallowing difficulties?' The Visual Analogue Scale (VAS) will be adopted to measure the degree of swallowing difficulties.
Change in the levels of sensation of pressure on soft tissue | T1: after 24 hours; T2: on the 7th day; T3: on the 15th day; T4: after 1 month; T5: after 4 months
  The degree of any sense of pressure in soft tissue that patients feel will be determined using their answers to the following question (question 04):
  ' What is the degree of any sense of pressure in soft tissue? ' The Visual Analogue Scale (VAS) will be adopted to measure the degree of any sense of pressure in soft tissue.

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Rabah, DDS,MSc, Principal Investigator — Specialist and Clinical Lecturer, Department of Orthodontics, University of Damascus; Heba M Al-Ibrahim, DDS,MSc, Principal Investigator — Specialist and Clinical Lecturer, Department of Orthodontics, University of Damascus; Mohammad Y Hajeer, DDS,MSc,PhD, Study Chair — Professor of Orthodontics, University of Damascus Dental School, Damascus, Syria; Rashad M.T. Murad, DDS,MSc,PhD, Study Chair — Professor of Pharmaceutics, University of Damascus, Faculty of Pharmacology, Damascus, Syria.
Locations (1):
- University of Damascus, Damascus, Syria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Saleh M, Hajeer MY, Al-Jundi A. Assessment of pain and discomfort during early orthodontic treatment of skeletal Class III malocclusion using the Removable Mandibular Retractor Appliance. Eur J Paediatr Dent. 2013 Jun;14(2):119-24. PMID 23758461
- [Background] Halicioglu K, Kiki A, Yavuz I. Subjective symptoms of RME patients treated with three different screw activation protocols: a randomised clinical trial. Aust Orthod J. 2012 Nov;28(2):225-31. PMID 23304972
- [Background] Feldmann I, Bazargani F. Pain and discomfort during the first week of rapid maxillary expansion (RME) using two different RME appliances: A randomized controlled trial. Angle Orthod. 2017 May;87(3):391-396. doi: 10.2319/091216-686.1. Epub 2016 Dec 28. PMID 28029266
- [Background] Ugolini A, Cossellu G, Farronato M, Silvestrini-Biavati A, Lanteri V. A multicenter, prospective, randomized trial of pain and discomfort during maxillary expansion: Leaf expander versus hyrax expander. Int J Paediatr Dent. 2020 Jul;30(4):421-428. doi: 10.1111/ipd.12612. Epub 2020 Jan 20. PMID 31894603
- [Background] De Felippe NL, Da Silveira AC, Viana G, Smith B. Influence of palatal expanders on oral comfort, speech, and mastication. Am J Orthod Dentofacial Orthop. 2010 Jan;137(1):48-53. doi: 10.1016/j.ajodo.2008.01.023. PMID 20122430